CLINICAL TRIAL: NCT04379622
Title: Differences in Dietary Intake, Body Composition, Lifestyle and Various Cardiovascular Diseases Risk Factors Among Healthy and Active Vegetrians and Non Vegetarians
Brief Title: Diet, Body Composition, Lifestyle and Cardiovascular Health of Healthy and Active Adults From Slovenia
Acronym: SloLifestyle
Status: Completed | Type: Observational
Sponsor: Barbara Jakše s.p. (Other)
Responsible Party: Principal Investigator, Boštjan Jakše, PhD student of Nutrition, Barbara Jakše s.p.
Other Study IDs: KR4
Record Dates: First submitted 2020-05-05; First posted 2020-05-07 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Diet, Healthy; Body Weight; Time Restricted Feeding; Sleep; Cardiovascular Risk Factor; Motivation
MeSH Terms: conditions — Body Weight; Intermittent Fasting | interventions — Eating; Body Composition

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional

INTERVENTIONS:
Other: Dietary intake, body composition, lifestyle, and CVD risk factors — Dietary intake, body composition, lifestyle, and CVD risk factors

SUMMARY:
There is objective need to evaluate the differences in dietary intake (DI), body composition (BC), lifestyle (LS) and cardiovascular diseases (CVD) risk factors between healthy and active vegetarinas (VEG) and non vegetarians (non VEG) and references (according to gender).

The aim of this cross-sectional study for investigators is to document the potential differences in DI (non adjusted and adjusted), BC, LS and CVD risk factors between healthy and active VEG and non VEG, aged from 18 to 80 years, and to evaluated correlation between DI variables and CVD risk factors.

The study during the COVID-19 pandemic period will be self-reported. As variables the investigators will include the dietary intake, BC (body height, body weight, body mass index (BMI), body fat percentage (BF %)), lifestyle status (physical activity, daily seating, hygiene of sleep, socio-economic status, and motive for practicing chosen diet). The investigators will also record their maximum (lifetime) body weight, lipids (total-cholesterol, LDL-cholesterol, HDL-cholesterol, and triglycerides) and blood pressure (BP) status.

The investigators hypothesis are:

(H1): There are differences in DI and quality of the diet (compared with references).

(H2): There are differences in BC between the VEG in non VEG (according to gender).

(H3): The are no differences between in CVD risk factors between the VEG and non VEG (according to gender).

(H4): The are no differences in the effect of two intervals of time restricted feeding (i.e., 8-12 hours vs. 12-16 hours) within dietary pattern (according to gender).

DETAILED DESCRIPTION:
In the study investigators will voluntarily enroll health and active 200-400 participants within inclusion/exclusion criteria that are willing to participate in the study. Investigators anticipate that for this number of adults (aged 18-80 years) will require approx. 10-20.000 invited candidates, of both sexes.

The methods to be used are standardized food frequency questionnaire (FFQ) that is sensible for different dietary patterns (to analyzed the daily dietary intake, for conventional component the investigators will use Dietplan7 Pro dietary assessment software (Forestield Software Limited, Horsham, UK), while for dietary supplements the investigators will use Res Pons d.o.o. servises, company that professionally manages a database with all dietary supplements and medicine products available on the Slovenian market.

BC status the investigators will use self-reported data from bioimpedance body composition monitor (Tanita, Tokyo, Japan), for basic anthropometric status the investigators will use medically approved body weight scale and body gauge (in the medical centers; body height, body weight, and BMI), and for lifestyle status the investigators will use three standardized questionnaires for: (1) habitual and organized physical activity, and the frequency of sitting (IPAQ-long), (2) quality of sleep (PSQI), and (3) socio-demographic, economic status adopted by Slovenian NIH.

Additionally, with added questionnaire the investigators will assessed the motives for VEG and non VEG dietary pattern. Investigators will record the participants maximum (lifetime) body weight (and therefore maximum BMI), and used self-reported CVD biochemistry results, measured in a standard and comparable method (plasma lipids, BP) in national medical centers.

ELIGIBILITY:
Inclusion Criteria:

* Health and active
* At least one year on same dietary pattern
* Signed informed consent to participate in the study
* Measured body composition status within last 90 days in Tanita body composition anayzer
* Measured values (annual or initiative examination report) of lipids and blood pressure

Exclusion Criteria:

* Major musculoskeletal restrictions
* Pregnant and lactating woman
* Currently competitive or top level athletes
* Current use of drugs for measured blood markers (lipids and blood pressure)
* Active common chronic diseases (i.e., cancer, CVD, autoimmune diseases ect.)
* Lost 5 kg or more within last year

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy and active Slovenian adults, without body mass index (BMI) limitation.
Sampling Method: Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2020-05-22 (Actual); Primary Completion 2020-08-05 (Actual); Study Completion 2020-08-05 (Actual)

PRIMARY OUTCOMES:
Body weight status | Cross-sectional (April-June 2020)
  Body weight measured with medically approved weighing scale
Height status | Cross-sectional (April-June 2020)
  Height status measured with medically approved weighing scale with height rod
Body mass index (BMI) status | Cross-sectional (April-June 2020)
  Measured weight and height will be combined to report BMI in kg/m2
Fat tissue mass status | Cross-sectional (April-June 2020)
  Fat tissue mass measured with bioimpedance analysis
Dietary intake status | Cross-sectional (May-June 2020)
  Dietary intake measured by food frequency questionnaire
Serum cholesterol status | Cross-sectional (May 2019-June 2020)
  Serum total cholesterol concentration
Oxidized Low Density Lipoprotein (LDL)-cholesterol status | Cross-sectional (May 2019-June 2020)
  Serum concentration of oxidized LDL-cholesterol
Serum HDL cholesterol status | Cross-sectional (May 2019-June 2020)
  Serum HDL cholesterol concentration
Serum triglyceride status | Cross-sectional (May 2019-June 2020)
  Serum triglyceride concentrations
Blood pressure status | Cross-sectional (May 2019-June 2020)
  Blood pressure status (systolic and diastolic)

SECONDARY OUTCOMES:
Socio-economic and demographic status | Cross-sectional (May-June 2020)
  Socio-economic and demographic status measured using Nutritional behaviours of adults Slovenians from the point of of health prevention questionnaire (Slovenian National Institute of Health)
Physical activity status | Cross-sectional (May-June 2020)
  Physical activity status measured by The International Physical Activity Questionnaires
Sleep status | Cross-sectional (May-June 2020)
  Sleep status measured with The Pittsburgh Sleep Quality Index
Motives for dietary pattern status | Cross-sectional (May-June 2020)
  Motives for dietary pattern status measured by investigators questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Boštjan Jakše, Principal Investigator — Barbara Jakše s.p.; Stanislav Pinter, PhD, Study Chair — University of Ljubljana
Locations (1):
- PDP Spodnje Črnuče, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] De Keyzer W, Dekkers A, Van Vlaslaer V, Ottevaere C, Van Oyen H, De Henauw S, Huybrechts I. Relative validity of a short qualitative food frequency questionnaire for use in food consumption surveys. Eur J Public Health. 2013 Oct;23(5):737-42. doi: 10.1093/eurpub/cks096. Epub 2012 Jul 26. PMID 22843611
- [Background] Hagstromer M, Oja P, Sjostrom M. The International Physical Activity Questionnaire (IPAQ): a study of concurrent and construct validity. Public Health Nutr. 2006 Sep;9(6):755-62. doi: 10.1079/phn2005898. PMID 16925881
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Fidler Mis N, Braegger C, Bronsky J, Campoy C, Domellof M, Embleton ND, Hojsak I, Hulst J, Indrio F, Lapillonne A, Mihatsch W, Molgaard C, Vora R, Fewtrell M; ESPGHAN Committee on Nutrition:. Sugar in Infants, Children and Adolescents: A Position Paper of the European Society for Paediatric Gastroenterology, Hepatology and Nutrition Committee on Nutrition. J Pediatr Gastroenterol Nutr. 2017 Dec;65(6):681-696. doi: 10.1097/MPG.0000000000001733. PMID 28922262
- [Derived] Jakse B, Jakse B, Godnov U, Pinter S. Nutritional, Cardiovascular Health and Lifestyle Status of 'Health Conscious' Adult Vegans and Non-Vegans from Slovenia: A Cross-Sectional Self-Reported Survey. Int J Environ Res Public Health. 2021 Jun 2;18(11):5968. doi: 10.3390/ijerph18115968. PMID 34199550
- See also: Forestfield Software Ltd. Forestfield Software - Dietplan — http://www.foresoft.co.uk/
- See also: NIJZ with partners (2019). — http://www.nijz.si/sl/podatki/nacionalna-raziskava-o-zdravju-in-zdravstvenem-varstvu-ehis-2019.
- See also: Guideline: sugars intake for adults and children — https://www.who.int/publications-detail/9789241549028
- See also: German Nutrition Society, Austrian Nutrition Society, Swiss Society of Nutrition Research, the S. A. for N. (2018). 3. Ergaenzlieferung D-A-CH Referenzwerte für die Nährstoffzufuhr [Reference Values for Nutrient Intake] (4th ed). — https://www.dge.de/wissenschaft/referenzwerte/
- See also: ResPons (2020) Pretehtajte prehranska dopolnila — https://pretehtajte.si/